CLINICAL TRIAL: NCT04661020
Title: Clinical Trial for the Safety and Efficacy of CD19 CAR-T Therapy for Patients With B-cell Non-Hodgkin's Lymphoma
Brief Title: CD19 CAR-T Therapy for Patients With B-cell Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19-003
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Non-hodgkin Lymphoma,B Cell
Keywords: Non Hodgkin Lymphoma; CAR T-cell therapy; CD19
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of CD19 CAR T-cells (Experimental)
  Interventions: Drug: CD19 CAR-T cells

INTERVENTIONS:
Drug: CD19 CAR-T cells — Each subject receive CD19 CAR T-cells by intravenous infusion
  Other Names: CD19 CAR-T cells injection

SUMMARY:
A Study of CD19 CAR-T Therapy for Patients With B-cell Non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for patients with CD19+ non-Hodgkin's lymphoma. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. 36 patients will be enrolled. Primary objective is to explore the safety, main consideration is dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age no less than 18, no gender limit;
2. Histologically confirmed diagnosis of HGBCL（HGBCL-NOS、HGBCL involving combined rearrangements of MYC, bcl-2 and bcl-6）DLBCL、not otherwise specified and IPI≥3;
3. Newly diagnosed B-NHL, unwilling to receive RCHOP first- or second-line chemotherapy, but willing to receive targeted drugs (such as a regimen consisting of CD20 monoclonal antibody，lenalidomide and Brutons tyrosine kinase inhibitor for two courses) as preconditioning regimens for CAR-T cell therapy;
4. Patients with PR or SD efficacy evaluated by PET-CT after two courses of tumor reduction therapy;
5. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit of normal, creatinine ≤ 176.8 umol/L;
6. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥50%;
7. No active infection in the lungs, blood oxygen saturation in indoor air is ≥ 92%;
8. Estimated survival time ≥ 3 months;
9. ECOG performance status 0 to 2;
10. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular, hemorrhagic diseases;
2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
3. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
4. Active infection of hepatitis B virus or hepatitis C virus;
5. Previously treated with any CAR-T cell product or other genetically modified T cell therapies;
6. Insufficient amplification capacity in response to CD3 / CD28 co-stimulus signal (<5 times) ;
7. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl;
8. Other uncontrolled diseases that were not suitable for this trial;
9. Patients with HIV infection;
10. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CD19 targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after CD19 targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
B-cell Non-Hodgkin's Lymphoma (B-NHL), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi) at Month 6, 12, 18 and 24
B-NHL, Overall survival (OS) | Up to 2 years after CD19 CAR-T cells infusion
  From the first infusion of CD19 CAR-T cells to death or the last visit
B-NHL, Event-free survival (EFS) | Up to 2 years after CD19 CAR-T cells infusion
  From the first infusion of CD19 CAR-T cells to the occurrence of any event, including death, relapse or generelapse,disease progression (any one occurs first), and the last visit
Quality of life(EORTC QLQ-C30) Core 30 (EORTC QLQ-C30) | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life QuestionnaireCore 30 (EORTC QLQ-C30) scale [For item1-28: max score: 112, min score: 28, higher scores mean a betteroutcome; for item 28-29: max score: 14, min score: 2, higher scores mean a worse outcome] to measure Quality of lifeat Baseline, Month 1, 3, 6, 9 and 12
Activities of Daily Living (ADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Activities of Daily Living (ADL) scale (Barthel Index) [max score: 100, min score: 0, higher scoresmean a better outcome] at Baseline, Month 1, 3, 6, 9 and 12
Instrumental Activities of Daily Living (IADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Instrumental Activities of Daily Living (IADL) scale [max score: 56, min score: 14, higher scores mean aworse outcome] at Baseline, Month 1, 3, 6, 9 and 12
Hospital Anxiety and Depression Scale (HADS) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Hospital Anxiety and Depression Scale (HADS) [max score: 42, min score: 0, higher scores mean aworse outcome] at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No